CLINICAL TRIAL: NCT05340933
Title: Speech and Voice As Biomarkers of Physiological Status in Patients with Respiratory Diseases: Proof of Concept in Acute Respiratory Disease Managed in a Pulmonary Hospital
Brief Title: Voice, Dyspnea and Acute Respiratory Failure
Acronym: LocuPnée-H
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: study discontinued
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: APHP211210
Record Dates: First submitted 2022-01-10; First posted 2022-04-22 (Actual); Last update posted 2024-10-02 (Actual); Status verified 2024-09

CONDITIONS: Acute Respiratory Diseases
Keywords: Acute respiratory failure; pneumonia; Chronic obstructive pulmonary desease; exacerbation; COVID-19 pneumonia; dyspnea; speech, voice analysis
MeSH Terms: conditions — Pneumonia; Dyspnea; Speech

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Arm 1 (Experimental): intervention correspond to the voice registration
  Interventions: Other: Voice registration

INTERVENTIONS:
Other: Voice registration — Voice registration

SUMMARY:
Breathing is an automatic vital function that has the peculiarity of being controllable voluntary for actions other than breathing. Speech production is a characteristic example of use of the respiratory system for nonrespiratory purposes. A healthy respiratory system is necessary for speech to be adequately produced and modulated. In patients with respiratory diseases, it becomes difficult to interfere with an automatic control of breathing that is intensely active to compensate for the respiratory deficience. Speech production is impeded, and, reciprocally, speech can generate dyspnea. This study explores the hypothesis that longitudinal changes in speech characteristics will parallel the clinical evolution of acute respiratory episodes. The aim is to validate such changes as prognostic indicators, in the perspective of future telemedicine applications. The hypothesis tested is that of an association between :

* vocal abnormalities at inclusion (assessed in relation to known data within a normal population (database of holy subjects already constituted) and the initial clinical severity (assessed according to the usual clinical and gasometric criteria):
* the evolution of vocal abnormalities during the stay and the clinical evolution.

DETAILED DESCRIPTION:
In the conceptual framework describe in the "brief summary" section of this document, this observational longitudinal monocentric study will include consecutive patients admitted in a specialised respiratory medicine ward for acute respiratory episodes. Any such episode will be considered be it "de novo" or complicating an underlying chronic respiratory disease. Vocal recordings will be performed daily, and will be analysed according to standard in the fields. Clinical parameters will also be recorded daily (vital signs, treatment intensity, outcome -including requirement for treatment intensification, transfer to the ICU, death, discharge to rehabilitation facility, discharge to home). The clinical follow-up and the vocal follow-up will be confronted to determine if voice analysis has an intrinsic prognostic value, alone, or in combination with clinical signs.

ELIGIBILITY:
Inclusion Criteria:

* patients hospitalised in the Pitié-Salpêtrière Pneumology Department with an acute respiratory illness (pneumonia of any cause, COVID pneumonia depending on the epidemic context, COPD decompensation, etc);
* whose condition allows conversational exchanges with the nursing staff within the framework of usual care;
* adults, not protected;
* understand and speak French fluently;
* affiliated to the social security system;
* having read and understood the information leaflet;
* do not object to the use of their data;

Exclusion Criteria:

* a clinical condition on admission that is too severe to allow the patient to answer the usual questions of the anamnestic and clinical examination
* patients with uncorrected hearing problems
* patients with neurological, otorhinolaryngological or psychiatric pathology

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2025-06-01 (Estimated); Primary Completion 2026-02-01 (Estimated); Study Completion 2026-09-01 (Estimated)

PRIMARY OUTCOMES:
Characterize voice analysis as a biomarker of respiratory status and its evolution in patients hospitalized in pneumology using machine learning algorithmshospitalized in pneumology | 1 month
  machine learning algorithms trained on the audio database obtained from patients discussion with medical staff. Voice parameters: respiratory rythms and intensity, and articulatory performances, will be extracted from voice recording, combined and analysed by the algorithms.

SECONDARY OUTCOMES:
Correlation of the used of algorithms based on voice and medical diagnosis. | 1 month
  Medical diagnosis based on physiological parameters (heart rate (bpm) ; oxygen saturation (%) ; respiratory rate (cycle/min)) will be carried out in the routine care and correlated with the algorythms results.

CONTACTS AND LOCATIONS:
Overall Officials: Thomas SIMILOWSKI, MD, PhD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Departement of Respiratory Medicine , Pitié-Salpêtrière Hospital, Paris, France, France